CLINICAL TRIAL: NCT06486987
Title: Efficacy of Constraint Induced Movement Therapy Delivered by Tele-Video for Children With Hemiplegic Cerebral Palsy
Brief Title: CHAMP T 2 Pilot of CIMT by Tele-Video
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Warren Lo (Other)
Collaborators: Ohio State University (Other); Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor-Investigator, Warren Lo, Clinical Professor, Pediatrics and Neurology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004128
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hemiplegic Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Participants with hemiplegic cerebral palsy will be treated with constraint induced movement therapy with the therapist participating by televideo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): This is a single arm in an open label pre- post-treatment design to estimate effect size of the intervention
  Interventions: Other: Constraint induced movement therapy delivered by televideo

INTERVENTIONS:
Other: Constraint induced movement therapy delivered by televideo — In-home Constraint induced movement therapy delivered by a therapist participating by televideo

SUMMARY:
The CHAMP-T2 study is a pilot test of the efficacy of constraint induced movement therapy (CIMT) when delivered by tele-video in the child's home or home-like environment. This study will examine the pre-, post-intervention function a hemiparetic limb in children who have hemiplegic cerebral palsy. The purpose is to provide an effect size estimate that will inform the design of a future study that will compare tele-delivered CIMT with usual and customary care.

DETAILED DESCRIPTION:
The CHAMP-T2 study is a pilot study of the efficacy of constraint induced movement therapy (CIMT) when delivered by tele-video in the child's home or home-like environment. This study will examine the pre-, post-intervention function of the paretic limb in children who have hemiplegic cerebral palsy. The purpose is to develop an effect size estimate that will inform the design of a future study that will compare tele-delivered CIMT with usual and customary care.

Primary Aim: To determine the effect of tele-delivered CIMT (CHAMP-T protocol) upon upper extremity (UE) motor function in school-aged children with post-stroke hemiparesis. The hypothesis is that the motor function of the paretic UE will improve significantly following tele-delivered CIMT.

The primary outcome will be the change in function of the impaired upper limb as measured by the Melbourne Assessment of Unilateral Upper Limb Function (MAUULF) (16) The secondary outcome will be the use of the affected limb in bilateral function as assessed with the Assisting Hand Assessment (AHA),(17) a well-established measure of an impaired upper limb in bilateral activities that is validated in children ages 18 months to 18 years. The parents will report their observation of the function of the affected limb also at baseline and at the end of the 4-week intervention. The reporting will use the Pediatric Motor Activity Log (PMAL),(18) which is a published, validated measure that was included in the study team's prior studies.(1) Fidelity to the treatment protocol will be assessed by parents' logs of the number of hours of treatment intervention the child undergoes, the recorded hours that the child wears the splint, and review of the recorded video sessions. Parent-therapist communication will be assessed by the Parent-Therapist information exchange tool. Factors affecting treatment delivery, including obstacles and barriers to task performance as well as supports that might assist performance in a larger clinical trial will be evaluated through semi-structured interviews and observations of treatment sessions with the parent and the treating therapist.

There will be a pre- and post-intervention assessment of the effect of tele-delivered CIMT delivered for 60 hrs over 4 weeks upon motor function of the paretic UE. After informed consent is obtained families will be asked to provide details regarding the child's medical history and diagnoses, previous treatments for cerebral palsy, and will be assessed for cerebral palsy severity.

The study will treat 10 children with hemiplegic cerebral palsy with the CHAMP-T2 protocol. Five families will be trained in- person by the therapists regarding basic principles of CIMT and how to use the televideo ensemble. Five families will receive the same training virtually. The CHAMP-T2 version of CIMT will be delivered 3 hours per day, 5 days per week, for 4 weeks by tele-delivery in the subject's home. The therapist will work with the parent by tele-video for 2 of the 3 hours to deliver the CIMT. The parent will work directly with the child without the therapist for a 3rd hour of each session. The children will wear the immobilization splint continuously each day up to 90% of the waking hours during the CIMT intervention period of 4 weeks.

The children will have UE motor function assessment at baseline and immediately post-treatment performed by blinded assessors. The parents, patients, and treating therapists will not be blinded.

After enrollment, a baseline assessment of motor function will be performed at the study center. For five children, the therapist then will travel to the child's home for 2 days of in-person training of the parent in the principles of CIMT and in the use of the iPad-Kubi Robot device. For the remaining five children the training will be performed by video. In the treatment phase of the study, the therapist will lead each therapy session by video for the first and third hours of the intervention. The second hour the parent will deliver the CHAMP-T2 intervention without the therapist on-line. During the therapist participation they will integrate parent coaching in the sessions to increase parent engagement and confidence with their delivery of the intervention. Video will be streamed live and recorded. Parent training and coaching will incorporate key elements (observation, action, reflection, feedback, and joint planning) (19) along with developing shared goal setting, problem solving and provision of feedback, education.

Fidelity to the treatment protocol will be assessed by parents' logs of the number of hours of treatment intervention the child undergoes, the recorded hours that the child wears the splint, and review of the recorded video sessions. Parent-therapist communication will be assessed by the Parent-Therapist information exchange tool. Factors affecting treatment delivery, including obstacles and barriers to task performance as well as supports will be evaluated through semi-structured interviews and observations of treatment sessions with the parent and the treating therapist. Parents will complete the Accessibility Intervention, Feasibility Intervention, and Intervention Appropriateness Measures (AIM, IAM, and FIM) to evaluate the treatment protocol and the Usefulness, Usability, and Desirability (UUD) measures to assess the study technology.

ELIGIBILITY:
Inclusion Criteria:

* Children who have hemiplegic cerebral palsy, ages 4-10;
* hemiparesis ranging from Manual Ability Classification System (MACS) I to MACS IV;
* live within a 1.5 hour distance from therapists' worksites at the Ohio State University Wexner Medical Center in Columbus, Ohio, or the Fralin Biomedical Research Institute in Roanoke, Virginia;
* are willing to travel to these sites for two in-person assessments.

Exclusion Criteria:

* Previous high dose CIMT (defined as CIMT given 2 hrs per day for 10 days) in the 6 months preceding baseline assessment;
* Treatment with botulinum toxin for spasticity in the 3 months preceding baseline assessment;
* Surgery for spasticity in the 6 months preceding baseline assessment;
* Medically unstable and unable to participate in the treatment intervention;
* Child is behaviorally or cognitively impaired so unable to participate in the treatment intervention;
* Family unable to participate in tele-delivery of CIMT 5 days a week for 4 weeks;
* the caregiver available at child's treatment site during treatment times is unable to communicate with the treating therapist.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Melbourne Assessment of Unilateral Upper Limb Function | At baseline pre-treatment and at the end of the 4-week intervention
  Measures function of the impaired upper limb

SECONDARY OUTCOMES:
Assisting Hand Assessment | At baseline pre-treatment and at the end of the 4-week intervention
  Measures function of the impaired upper limb in bilateral upper limb functions
Pediatric Motor Activity Log | At baseline pre-treatment and at the end of the 4-week intervention
  Parent reported assessment of upper limb motor activity
Fidelity to treatment protocol | During 4 weeks of intervention
  Parent logs of numbers of hour of treatment and hours the child wears constraint

CONTACTS AND LOCATIONS:
Overall Officials: Warren Lo, MD, Principal Investigator — Nationwide Children's Hospital
Locations (2):
- United States (2):
  - The Ohio State University School of Health and Rehabilitation Sciences, Columbus, Ohio
  - Virginia Tech-Fralin Biomedical Research Institute, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No
For this small pilot study we do not anticipate sharing individual participant data because of the difficulty of maintain subject confidentiality

REFERENCES:
- [Background] Ramey SL, DeLuca SC, Stevenson RD, Conaway M, Darragh AR, Lo W; CHAMP. Constraint-Induced Movement Therapy for Cerebral Palsy: A Randomized Trial. Pediatrics. 2021 Nov;148(5):e2020033878. doi: 10.1542/peds.2020-033878. Epub 2021 Oct 14. PMID 34649982